CLINICAL TRIAL: NCT06810713
Title: Evaluation of a Training for Healthcare Providers in Supporting Men Experiencing Suicidal Ideation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0536
Record Dates: First submitted 2025-01-22; First posted 2025-02-05 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gatekeeper training (e-learning) (Experimental): Participants in this group (all participants) are asked to complete a questionnaire and then receive access to the online training (e-learning), after which they were asked to complete another questionnaire. In case a participant does not complete the post-test, a reminder will be sent via e-mail three days later.
  Interventions: Behavioral: Gatekeeper training (e-learning)

INTERVENTIONS:
Behavioral: Gatekeeper training (e-learning) — This training supplements existing modules for healthcare providers working with individuals experiencing suicidal thoughts (https://sp-reflex.zelfmoord1813.be/e-learning).
  Specific information on working with men will be added:
  * Information on suicidality among men and the importance of gender-sensitive care.
  * Guidance on recognizing signs of suicidality in men and understanding gender differences in suicide-related communication.
  * Insights into the impact of gender norms and socialization on suicidality and help-seeking behavior in men experiencing suicidal thoughts.
  * Awareness of providers' own gender biases and the influence of societal gender norms in treating men with suicidal ideation.
  * Recommendations for engaging men in treatment, with specific guidance on language and approaches for interacting with men who have suicidal thoughts.
  Additionally, the e-learning will a model psychoeducation about the role of norms for men experiencing suicidal ideation.

SUMMARY:
The primary objective of this study is to assess how healthcare providers perceive and evaluate the developed e-learning. The findings will inform potential adjustments to enhance the e-learning as needed.

DETAILED DESCRIPTION:
In a previous study (BUN: B6702024000090), the authors focused on identifying barriers and needs among adult men experiencing suicidal thoughts and their healthcare providers. Findings from this needs assessment indicate a demand for a training (e-learning) to equip healthcare providers with strategies for working effectively with men experiencing suicidal ideation. Additionally, the assessment among individuals with suicidal ideation identified several key recommendations and considerations which healthcare providers should incorporate into their practice. Therefore, an e-learning was developed with integrated psycho-education and the primary objective of this study is to assess how healthcare providers perceive and evaluate the developed e-learning. The findings will inform potential adjustments to enhance the e-learning as needed.

Participants will be recruited through announcements on the Flemish suicide prevention portal website (www.zelfmoord1813.be) and websites of relevant partners (i.e. VVKP, VVP, Gezond Leven, Psyché, Vivel, Logo's, CGG-SP, Domus Medica,…), as well as via social media (mainly Linkedin, Instagram and Facebook) and newsletters of the Flemish Centre of Expertise in Suicide Prevention and its relevant partner organizations.

Individuals interested in participating will be directed to register online through REDCap, where they will review and approve an informed consent form.After providing informed consent, participants will be asked to provide their email address.

The email address will be used solely for the following purposes:

- Sending a reminder to complete the post-test questionnaire three days later. Once consent is provided, participants will be directed to the online pre-test questionnaire (see Table 1), which takes approximately 10 minutes to complete. Following the pre-test, participants will be directed to the e-learning module, which requires 30-60 minutes. At the end of the e-learning, healthcare providers will be asked to complete the post-test questionnaire, which is estimated to take 15 minutes. In case a participant does not complete the post-test, a reminder will be sent via e-mail three days later.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (e.g. GP's, psychiatrists, medical doctors, psychologists, psychotherapists, and nurses working in healthcare)
* ≥18y/o
* Access to a smartphone, tablet, or computer with internet connection and proficiency in Dutch

Exclusion Criteria:

* Does not meet the specified inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Competencies related to working with male clients (self-efficacy) | Change from Baseline (before e-learning) to post-test (immediatly after e-learning of 30-60 minutes); assessed up to 3 days after pre-test
  Adaptation of the Engaging Men in Therapy Scale (EMITS): scale of 13 items to be rated on a scale from 1 (strongly disagree) to 5 (strongly agree), resulting in a total score of 13-65. Higher scores indicating higher self-reported competency for engaging with male clients.
  The adapted version consists of 8 items, as not all aspects of the original questionnaire are included in the evaluated e-learning.
Evaluation of the training | Post-test (immediatly after e-learning of 30-60 minutes), up to 3 days after pre-test
  self-developed questionnaire: score on a scale of 1 (not good at all) to 10 (Excellent); 10 evaluation statements to be rated on a scale of 1 (totally disagree) to 5 (totally agree); 9 open questions; one question about the length of the e-learning (too short, too long or just fine)

SECONDARY OUTCOMES:
self-efficacy | Change from Baseline (before e-learning) to post-test (immediatly after e-learning of 30-60 minutes); assessed up to 3 days after pre-test
  self-efficacy in working with men experiencing suicidal ideation: 2 questions on self-rated competence in recognizing and inquiring about suicide (1), discussing suicidal ideation withmen (2)to be rated on a 5-point scale (Not competent at all to very competent).

OTHER OUTCOMES:
Socio-demographic variables | Baseline
  Gender and age
Work situation | Baseline
  Self-developed questionnaire: Type of healthcare provider, current work place, experience, previous training in suicide prevention
Experience with men with suicidal thoughts | Baseline
  one question about experience with men with suicidal thoughts

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seidler ZE, Wilson MJ, Benakovic R, Mackinnon A, Oliffe JL, Ogrodniczuk JS, Kealy D, Owen J, Pirkis J, Mihalopoulos C, Le LK, Rice SM. A randomized wait-list controlled trial of Men in Mind: Enhancing mental health practitioners' self-rated clinical competencies to work with men. Am Psychol. 2024 Apr;79(3):423-436. doi: 10.1037/amp0001242. Epub 2023 Nov 27. PMID 38010768